CLINICAL TRIAL: NCT02539706
Title: The Impact of the Menstrual Cycle on Injection Pain of Rocuronium
Brief Title: Menstrual Cycle on Injection Pain of Rocuronium
Acronym: MENS
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Aydin Adnan Menderes University (Other)
Responsible Party: Principal Investigator, SİNAN YILMAZ, Associate Professor, Aydin Adnan Menderes University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Diagnostic
Other Study IDs: sinan
Record Dates: First submitted 2015-09-01; First posted 2015-09-03 (Estimated); Last update posted 2017-11-29 (Actual); Status verified 2017-11

CONDITIONS: Pain, Menstrual
MeSH Terms: conditions — Dysmenorrhea | interventions — Rocuronium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Follıcular group (Experimental): patients at days 8 to 14 of the menstrual cycle were considered to be at the follicular phase and Rocuronium 0,6mg/kg intravenous rocuronium was applied.
  Interventions: Drug: Rocuronium 0,6mg/kg
- Luteal group (Active Comparator): patients at days 18 to 24 of the menstrual cycle were considered to be at the luteal phase and Rocuronium 0,6mg/kg intravenous rocuronium was applied.
  Interventions: Drug: Rocuronium 0,6mg/kg

INTERVENTIONS:
Drug: Rocuronium 0,6mg/kg — patients at days 8 to 14 of the menstrual cycle were considered to be at the follicular phase and Rocuronium 0,6mg/kg intravenous was applied
  Other Names: esmeron
  Arms: Follıcular group
Drug: Rocuronium 0,6mg/kg — patients at days 18 to 24 of the menstrual cycle were considered to be at the luteal phase and Rocuronium 0,6mg/kg intravenous rocuronium was applied
  Other Names: esmeron
  Arms: Luteal group

SUMMARY:
This study evaluates the effects of rocuronium injection pain to menstrual cycle phases.Half of participants will receive follicular phase, while the other half will receive luteal phase.

DETAILED DESCRIPTION:
Menstrual period includes a spectrum of emotional and somatic symptoms observed in luteal phase of menstrual cycle, which are disappeared after menstruation.

During menstrual cycle, fluctuation in sexual hormones results in attitude change and alteration in pain perception.

Different studies reported some interactions between sex hormones and central nervous system, which might be linked to activity of serotonin and beta-endorphin in the brain.

Pain perception differs during menstrual cycle.

It has been recommended that estrogens might have an influence on somatic sensory process.

Some studies reported a significant effect of pain sensitivity with higher levels of progesterone and some other studies reported similar patterns for pain perception.

There are reports of more complaint of pain in luteal phase of menstruation, which is suggested as the reason for functional changes in women during menstrual cycle.

ELIGIBILITY:
Inclusion Criteria:

* American Society of Anesthesiology Classification (ASA) I-II
* 18-45 years
* Regular menstrual cycle

Exclusion Criteria:

* Irregular menstrual cycles
* Patients receiving hormones or drugs affecting the ovulatory cycle
* Amenorrhea
* Pregnancy
* Climacteric patients

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2014-01-06 (Actual); Primary Completion 2015-09-06 (Actual); Study Completion 2015-10-06 (Actual)

PRIMARY OUTCOMES:
Pain measure | 10 second
  Tracheal intubating dose of 0.6 mg/kg of rocuronium at room temperature was injected over 10 -15 s. The patients were observed immediately if they had pain in the arm, and the response was assessed. Withdrawal movements were also assessed and scored as follows: no movements = 0, movement limited to hand = 1, movement limited to the forearm including the elbow joint = 2, and movement of the upper arm including the shoulder joint = 3

CONTACTS AND LOCATIONS:
Overall Officials: Adnan Menderes Univercity Medicine Faculty, Principal Investigator — Adnan Menderes University,Faculty of Medicine, Department of Anesthesia
Locations (1):
- Adnan Menderes University Training and Research Hospital, Aydin, Turkey (Türkiye)